CLINICAL TRIAL: NCT03514628
Title: Evaluation of Pre-hospital Use of a Valsalva Assist Devise (VAD) in the Emergency Treatment of Supraventricular Tachycardia (SVT). A Randomised Controlled Feasibility Trial [EVADE]
Brief Title: Evaluation of the Valsalva Assist Device to Treat SVT
Acronym: EVADE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Western Ambulance Service NHS Foundation Trust (Other)
Collaborators: Royal Devon and Exeter NHS Foundation Trust (Other); Academic Health Science Centres (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 238130
Record Dates: First submitted 2018-04-10; First posted 2018-05-02 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: SVT; Vagal Bradycardia; Emergencies
Keywords: Valsalva Manoeuvre; SVT; Valsalva Assist Device
MeSH Terms: conditions — Emergencies | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: 1:1 randomisation to VAD or standard care
Who Masked: Investigator, Outcomes Assessor
Masking Description: Data analysis and determination of primary outcome will be done blind to allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Valsalva Assist Device (VAD) (Experimental): Intervention is the use of Valsalva Assist Device (VAD) to deliver the Valsalva strain
  Interventions: Device: Valsalva Assist Device (VAD)
- Standard Care (Active Comparator): Intervention is the use of Standard technique to deliver Valsalva strain eg blowing on empty syringe
  Interventions: Other: Standard Care

INTERVENTIONS:
Other: Standard Care — The Valsalva strain will be produced using Standard Care techniques
  Arms: Standard Care
Device: Valsalva Assist Device (VAD) — Use of Valsalva Assist Device (VAD) to generate VM
  Arms: Valsalva Assist Device (VAD)

SUMMARY:
The Valsalva Assist Device (VAD) is a simple hand held device, designed to assist in the physical treatment of a common, fast heart rhythm disorder called supraventricular tachycardia (SVT).

This treatment, called the Valsalva manoeuvre (VM), is a safe, physical technique involving a forced exhalation against resistance (like that required to blow up a balloon). This causes a reflex slowing of the heart and can correct attacks of SVT (cardioversion). It is an internationally recommended initial treatment but previously has had a low success rate (5-27%) and patients often have to be taken to hospital for drug treatment.

Recent hospital research has demonstrated that a VM carried out using a certain level of strain pressure(40mmHg) measured with a blood pressure manometer, combined with a simple postural modification (the modified VM) gives a far better chance of success (43%) and avoids the need for drug treatment. More practical methods of generating this strain such as blowing on an empty syringe have been used but are unreliable. The Valsalva Assist Device (VAD) has been designed to provide the correct resistance and is packaged with instructions for the modified VM.

Attacks of SVT frequently occur without warning in otherwise healthy people. Patients are often initially seen by ambulance staff and so the use of the VAD therefore represents an opportunity to provide ambulance clinicians with instructions for the modified VM and a means to deliver the correct strain in one, easy to use device.

The investigators plan to test use of the device in patients with an attack of SVT and attended by paramedics or other pre-hospital practitioner, compared to current recommended practice. This project will provide important feasibility and recruitment data for a definitive trial, assessing the performance of the VAD on SVT cardioversion and conveyance (transfer to hospital) rates.

DETAILED DESCRIPTION:
The investigators plan to conduct a pragmatic, randomised controlled trial of the use of the Valsalva Assist Device (VAD) versus standard care to treat SVT delivered by ambulance clinicians.

Ambulance clinicians within South West Ambulance Service Foundation Trust (SWASFT) will be invited to help deliver this study by becoming recruiting practitioners. All participating ambulance clinicians will have specific trial training including an update of SVT management, use of the VAD and GCP training as needed. It is estimated a two month ambulance clinician recruitment period would enable approximately 80 clinicians to be enrolled.

Patients presenting with SVT to these trained participating ambulance clinicians will be screened according to the eligibility criteria during their initial clinical assessment over a 6-8 month concurrent recruitment period. This will include routine observations and recording of an ECG.

Eligible participants will be informed about the nature of SVT and the VM as the initial recommended treatment. They will then take part in a structured verbal consent process, witnessed by a second member of ambulance staff or nominated individual such as a relative or friend. They will be given a verbal explanation of the study and that the proposed treatment differs only in the method used to generate the Valsalva strain and that all other management is entirely as normal. It will be stressed that they are under no obligation to take part and that the method of producing the strain will be chosen at random on the opening of a box containing a simple device (VAD) or instructions advising usual practise such as blowing into a syringe.

These boxes will be indistinguishable and distributed to participating ambulance clinicians at random. Clinicians will carry one box at a time and restock by taking the next available lowest numbered box from their ambulance station when used. They will be closed with a tamper evident seal and not opened until the witness has confirmed the patient's verbal consent to take part and that the box's seal is intact.

Consenting participants will undergo a maximum of three Valsalva manoeuvres under direction of the treating crews according to training and allocation of device or standard care. All other treatment and subsequent clinical management will be according to national and local guidelines. This includes ongoing observations and ECGs as recorded on the ambulance electronic patient record (ePCR). Participants who remain in SVT will be conveyed to hospital as is standard practice. For participants whose SVT has cardioverted back to normal sinus rhythm, there is an excisting locally approved protocol for non-conveyance of well patients at the discretion of the treating ambulance clinician. This includes a plan for ongoing follow up by the patient's GP.

All participants will be given a written information sheet at a suitable time after pre-hospital treatment is complete. This will give further details of the research, contact details for the research team and clear instructions on how to withdraw from further participation or use of their data. Paramedics will also verbally confirm that participants are still willing to be included and ask if they would be happy to be contacted for a brief 5 minute telephone follow up call by a member of the research team to ask their views on the consent process and other trial procedures. Participants will also be offered the device or a syringe to take away depending on their allocation. The written advice will include reminder instructions on how to perform a VM themselves as SVT can recur and self treatment is recommended if patients would like to try this.

Screening and notification of recruitment will be taken from the ambulance electronic patient record (ePCR) which has a field to indicate involvement in a research program. Evidence of participation will also be collected by return or photo (on ePCR) of the opened, completed lid of the trial allocation box. All other data collection will as far as possible mirror normal procedures. Source and outcome data will also be taken from the ePCR. Primary outcome data (ECG) will be checked by an independent consultant emergency physician, blind to the patient's trial allocation. Where disagreement, arbiter (consultant cardiologist) assessment will be made and confirmed by independent outcome committee. No other routine trial follow up is planned. However, adverse events will be reported and followed up according to good clinical practice (GCP) principles.

Statistical analysis will be conducted on intention to treat basis blind to allocation. Recruitment and baseline cardioversion rates will enable subsequent sample size estimates to be made for the definitive trial grant application.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (above 17years)
* Presenting with SVT which the ambulance clinician identifies as being eligible for a vagal manoeuvre

Exclusion Criteria:

* Unable or unwilling to give informed verbal consent
* Unstable condition (systolic blood pressure (BP) < 90mmHg) [Increased risk of feeling or actually fainting with a VM which causes a transient fall in BP as a normal physiological response]
* Atrial fibrillation or atrial flutter on ECG [VM considered ineffective in these rhythms]
* Severe hypertension (systolic BP >220mmHg or diastolic BP >120mmHg) [Risk of further increase in BP at end of VM - a normal physiological response]
* Contraindication or inability to perform a modified Valsalva manoeuvre in the opinion of the practitioner. This will include but not limited to: Aortic stenosis, recent myocardial infarction, glaucoma, retinopathy and inability to perform a Valsalva manoeuvre, to lie flat or have legs lifted. [We will exclude all those that could conceivable come to any harm from performing a VM]
* Third trimester pregnancy [Lying flat can cause fainting in late pregnancy]
* Prisoners
* Previous inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Clinician recruitment | At study completion (after an 8 month recruitment period)
  A key measures for this pilot project will be the rate of ambulance clinician recruitment.
Participant recruitment | At study completion (after an 8 month recruitment period)
  The number of participants recruited to the trial

SECONDARY OUTCOMES:
Cardioversion rates | At study completion (after an 8 month recruitment period)
  The proportion of participants who are returned to sinus rhythm as determined by ambulance ECG after the VM. The primary outcome in the definitive study will be return to sinus rhythm after paramedic Valsalva manoeuvre attempts as determined by the treating ambulance clinician and confirmed by evidence from the ePCR such as 12 lead ECG s. This project will assess the feasibility of capturing this outcome measure.
Conveyance rates | At study completion (after an 8 month recruitment period)
  The proportion of participants who are conveyed to hospital. This will be an alternative primary outcome in the definitive study and so this project will also assess the feasibility of capturing this outcome measure.
Completeness of data | At study completion (after an 8 month recruitment period)
  The proportion of all data fields available and completed at the end of the study. Availability and completeness of all data

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Appelboam, MBBS, FRCEM, Principal Investigator — Royal Devon and Exeter NHS Foundation Trust
Locations (1):
- 29 Selected Ambulance Stations, Exeter, South West England, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Appelboam A, Green J, Ewings P, Black S; EVADE study SWASFT collaborators. Evaluation of pre-hospital use of a valsalva assist device in the emergency treatment of supraventricular tachycardia [EVADE]: a randomised controlled feasibility trial. Pilot Feasibility Stud. 2020 May 25;6:74. doi: 10.1186/s40814-020-00616-y. eCollection 2020. PMID 32509319